CLINICAL TRIAL: NCT03433521
Title: Observational Study of Spatio-Temporal Patterns of New Cases of Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: EO 100/2017_FJD-HRJC
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Spatio-Temporal Diagnostic Pattern
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Published data regarding the temporal pattern of AML are scarce and old. The greater knowledge of these neoplasias has made that their classification has been remarkable modified. Therefore, we consider relevant to carry out the present study as it would allow us to analyze the potential existence of a spatio-temporal pattern in the incidence of AML in Spain.

ELIGIBILITY:
Inclusion Criteria Patients with a first diagnostic of AML between 2004 and 2014.

.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Spanish population
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
AML diagnosis | 10 years
  Diagnosis of de-novo AML

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Investigacion Sanitaria Fundacion Jimenez Diaz, Madrid, Spain